CLINICAL TRIAL: NCT03592498
Title: Randomised Clinical Study to Evaluate the Use of Tilapia Skin (Oreochromis Niloticus), as an Occlusive Biological Dressing, in the Treatment of Burn Wounds
Brief Title: Study to Evaluate the Use of Tilapia Skin (Oreochromis Niloticus), in the Treatment of Burn Wounds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara (Other)
Responsible Party: Principal Investigator, Edmar Maciel Lima Júnior, MD, Plastic Surgeon, Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pele de tilápia
Record Dates: First submitted 2018-05-25; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Burns
Keywords: Burns; Wounds and Injuries; Biocompatible Materials; Nile Tilapia; Oreochromis niloticus.
MeSH Terms: conditions — Burns; Wounds and Injuries | interventions — Silver Sulfadiazine

STUDY DESIGN:
Intervention Model Description: Clinical study Phase II, pilot, open, monocentric and randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulfadiazine, Silver (Active Comparator): Intervention: Treatment with silver sulfadiazine ointment. Procedures: wound washing, application of silver sulfadiazine ointment, bandage covered with gauze and bandage. These patients undergone the change of dressings on alternate days.
  Interventions: Drug: Sulfadiazine, Silver
- Skin of Nile tilapia (Experimental): Intervention: treatment with skin of Nile tilapia (Oreochromis niloticus), as a biological occlusive dressing.
  Procedures: wound washing, application of tilapia skin and dressing with gauze and bandage. These dressings were changed if the skin of the tilapia was loose (not adhered).
  Interventions: Device: Skin of Nile tilapia

INTERVENTIONS:
Drug: Sulfadiazine, Silver — Application of silver sulfadiazine ointment, bandage covered with gauze and bandage.
  Arms: Sulfadiazine, Silver
Device: Skin of Nile tilapia — Application of skin of Nile tilapia (Oreochromis niloticus), as a biological occlusive dressing.
  Arms: Skin of Nile tilapia

SUMMARY:
Randomised Clinical Study to evaluate the efficacy of Nile tilapia (Oreochromis niloticus) skin as an occlusive biological dressing, in the treatment of humans burn wounds.

DETAILED DESCRIPTION:
This was a randomized, monocentric; open-label pilot clinical study conducted at the Dr. José Frota Institute's Burn Treatment Center, located in Fortaleza, Ceará, Brazil, from October 2016 to September 2017.

The study participants were recruited from the population of patients attending the Burning Treatment Center of the Dr. José Frota Institute. Were included female and male participants, age range greater than or equal to 18 and greater than or equal to 50 years old and who met the following criteria: presence of a dermatological wound caused by superficial second-degree burn with up to 20% of the body surface or deep second degree with area of 5 to 15% of the body surface; absence of previous treatment for the current burn and without other significant diseases that could impact their participation in the study. No study participants were known to have hypersensitivity to materials used in the study or to related compounds; history of serious adverse reactions; addiction to drugs, including alcohol; pregnancy and labor or miscarriage in the 12 weeks prior to the scheduled start of treatment.

The study was divided according to the depth and burned body surface area of the research participant:

Study A: Burning of 2nd Surface Degree with <10% of body surface area - Patients in outpatient care, within this group, the research participants were randomly assigned to the following treatment groups: active comparator (sulfadiazine, Silver) or experimental (skin of Nile tilapia).

Study B: 2nd Degree Burn with 10 to 20% body surface area - Inpatient, within this group, the research participants were randomly assigned to the following treatment groups: active comparator (sulfadiazine, Silver) or experimental (skin of Nile tilapia).

Study C: Deep 2nd Degree Burn with 5 to 15% body surface area - Inpatient, within this group, the research participants were randomly assigned to the following treatment groups: active comparator (sulfadiazine, Silver) or experimental (skin of Nile tilapia).

Interventions:

Participants were randomly assigned to the following treatments:

* Experimental intervention: use of the skin of Nile tilapia (Oreochromis niloticus), as a biological occlusive dressing;
* Active comparator intervention: Conventional treatment with silver sulfadiazine.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a dermatological wound caused by superficial second-degree burn with up to 20% of the body surface or deep second degree with area of 5 to 15% of the body surface;
* Absence of previous treatment for the current burn
* Without other significant diseases that could impact their participation in the study

Exclusion Criteria:

* Hypersensitivity to materials used in the study or to related compounds;
* History of serious adverse reactions;
* Addiction to drugs, including alcohol;
* Pregnancy
* Labor or miscarriage in the 12 weeks prior to the scheduled start of treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Number of days for complete re-epithelization in study A and B | Day 11
  Number of days until complete re-epithelialization observed by the evaluator
Number of days for complete re-epithelization in study C | Day 21
  Number of days until complete re-epithelialization observed by the evaluator
The number of dressings performed as needed in study A and B | Day 11
  Relation to the number of dressings performed in patients treated with Silver Sulfadiazine and Tilapia Skin throughout the treatment.
The number of dressings performed as needed in study C | Day 21
  Relation to the number of dressings performed in patients treated with Silver Sulfadiazine and Tilapia Skin throughout the treatment.
Amount of anesthetics or analgesics used throughout the treatment in study A and B | Day 11
  Use of anesthetics or analgesics required for the change of dressings performed throughout the treatment.
Amount of anesthetics or analgesics used throughout the treatment in study C | Day 21
  Use of anesthetics or analgesics required for the change of dressings performed throughout the treatment.

SECONDARY OUTCOMES:
Change in scale of pain by the Visual Analogue Scale | Day 1, 3, 5, 7, 9, 11, 15 and 30 (group A and B) and day 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25 and 40 (group C).
  The visual Analogue scale consists of assisting in the assessment of pain intensity in the patient, being an important instrument to verify the evolution of the patient during the treatment. In each visit, the patient was instructed to respond as he rated his pain through scores ranging 0 to 10, where 0 to 2 meant mild pain, 3 to 7 meant moderate pain and 8 to 10 meant severe pain.
Change in Global Clinical Impression Scale - Disease Severity (CGI-S) scores | Day 1, 3, 5, 7, 9, 11, 15 and 30 (group A and B) and day 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25 and 40 (group C).
  The evaluation of change in the scores of burn severity was performed by the physician during the study, using the global clinical impression scale - disease severity, which consistes of answering the following question - Considering your experience with this type of problem, what is the degree of severity of this patient's illness at the moment?? - Where, 0 means not evaluated, 1 - Much better, 2 - moderately better, 3 - Slightly better, 4 - unchanged, 5 - Slightly worse, 6 - Moderately worse and 7 - Much worse.
Change in Global Clinical Impression Scale - Disease Improvement (CGI-I) scores | Day 1, 3, 5, 7, 9, 11, 15 and 30 (group A and B) and day 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25 and 40 (group C).
  The evaluation of change in the scores of burn improvement was performed by the physician during the study, using the global clinical impression scale - disease improvement, which consists of answering the following question - Compared to the initial state, how is the patient at this time? - Where, 0 means Not evaluated, 1 - Much better, 2 - moderately better, 3 - Slightly better, 4 - unchanged, 5 - Slightly worse, 6 - Moderately worse and 7 - Much worse.
Change in patient global assessment scores | Day 1, 3, 5, 7, 9, 11, 15 and 30 (group A and B) and day 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25 and 40 (group C).
  The change in the patient burn-related symptoms was realized by answering the following question: Compared to the initial state, how is your disease-related symptoms at this time? - Where, 0 means much better, 1 - moderately better, 2 - Slightly better, 3 - unchanged, 4 - Slightly worse, 5 - Moderately worse and 6 - Much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisabete A Moraes, MD, Study Director — Clinical Pharmacology Unit, Drug Research and Development Center, Federal University of Ceara (UFC)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alves APNN, Lima Junior EM, Piccolo NS, de Miranda MJB, Lima Verde MEQ, Ferreira Junior AEC, de Barros Silva PG, Feitosa VP, de Bandeira TJPG, Mathor MB, de Moraes MO. Study of tensiometric properties, microbiological and collagen content in nile tilapia skin submitted to different sterilization methods. Cell Tissue Bank. 2018 Sep;19(3):373-382. doi: 10.1007/s10561-017-9681-y. Epub 2018 Jan 29. PMID 29380095
- [Derived] Lima Junior EM, De Moraes Filho MO, Costa BA, Rohleder AVP, Sales Rocha MB, Fechine FV, Forte AJ, Alves APNN, Silva Junior FR, Martins CB, Mathor MB, Moraes MEA. Innovative Burn Treatment Using Tilapia Skin as a Xenograft: A Phase II Randomized Controlled Trial. J Burn Care Res. 2020 May 2;41(3):585-592. doi: 10.1093/jbcr/irz205. PMID 31900475
- See also: Article about the tilapia skin — http://rbqueimaduras.org.br/details/341/pt-BR/uso-da-pele-de-tilapia--oreochromis-niloticus---como-curativo-biologico-oclusivo--no-tratamento-de-queimaduras
- See also: Article about the tilapia skin — http://periodicos.unichristus.edu.br/index.php/jhbs/article/view/767
- See also: Article about the tilapia skin — http://rbqueimaduras.org.br/details/263/pt-BR/avaliacao-microscopica--estudo-histoquimico-e-analise-de-propriedades-tensiometricas-da-pele-de-tilapia-do-nilo